CLINICAL TRIAL: NCT00054431
Title: Phase II Study of Imatinib Mesylate (Gleevec, STI-571) (NSC#716051) and Decitabine (5-AZA-2'-Deoxycitidine) (NSC#127716), in Chronic Myelogenous Leukemia in Accelerated and Blastic Phases
Brief Title: Imatinib Mesylate and Decitabine in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02516; MDA-ID-02205; N01CM62202 (NIH); CDR0000270678 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Childhood Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Relapsing Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Decitabine

ARMS (1):
- Treatment (imatinib mesylate, decitabine) (Experimental): Patients receive oral imatinib mesylate daily and decitabine IV over 1 hour daily, 5 days per week, for 2 consecutive weeks. Courses repeat every 4-6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Drug: decitabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving imatinib mesylate together with decitabine works in treating patients with accelerated or blast phase chronic myelogenous leukemia. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Giving imatinib mesylate together with decitabine may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the duration of response and response rate in patients with accelerated or blastic phase chronic myelogenous leukemia treated with imatinib mesylate and decitabine.

II. Determine the survival rate of patients treated with this regimen. III. Determine the toxicity of this regimen in these patients. IV. Determine the effects of this regimen on gene methylation in the leukemic cells of these patients.

OUTLINE: Patients are stratified according to prior exposure to imatinib mesylate (yes vs no).

Patients receive oral imatinib mesylate daily and decitabine IV over 1 hour daily, 5 days per week, for 2 consecutive weeks. Courses repeat every 4-6 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 20-80 patients (10-40 per stratum) will be accrued for this study within 20 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic myelogenous leukemia

  * Philadelphia chromosome positive by cytogenetics OR fluorescent in situ hybridization
  * Accelerated or non-lymphoid blastic phase
* Performance status - ECOG 0-2
* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 2 times ULN
* Creatinine less than 2.0 mg/dL
* Normal cardiac function
* No New York Heart Association class III or IV heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior decitabine
* At least 2 weeks since other prior chemotherapy (unless there is evidence of rapidly progressive disease) and recovered
* Concurrent hydroxyurea allowed during the first 2 courses of study therapy in patients with rapidly progressing disease
* Prior imatinib mesylate allowed

  * Patients who received at least 4 weeks of prior imatinib mesylate must have failed therapy, as evidenced by resistance after 8 weeks or disease progression
* No concurrent grapefruit or grapefruit juice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-01; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Complete and partial response | 6 months
Hematologic improvement | Up to 1 year
Duration of response | Date of documented response until relapse, assessed up to 4 years

SECONDARY OUTCOMES:
Toxicities, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Issa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States